CLINICAL TRIAL: NCT03992040
Title: Assessment of Medico-economic Relevance of Care of Polypathological Patients by a Reinforced Home Nursing Care Services (SSIAD)Device
Brief Title: Assessment of Medico-economic Relevance of Care of Polypathological Patients by a Reinforced Home Nursing Care Services (SSIAD) Device
Acronym: SSIADR
Status: Completed | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01188-49
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Polypathological Patient Having Obtained a Place in Home Nursing Care Services SSIAD by Medical Prescription
Keywords: Regional Public Health authorities (ARS) score; Reinforced Home Nursing Care Services (SSIADR)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reinforced SSIAD (SSIADR arm ): Reinforced Home Nursing Care Services: Patients with a score between 11 and 21 on the regional public health authorities (ARS) score.
  This arm will benefit from better coordination and delivery of care, which can reduce hospitalizations and visits to emergency departments
- Classic SSIAD (Control arm): Classic Home Nursing Care Services. For this arm, no direct benefit is expected since taking care, even for the heaviest patients, corresponds to current practice.

SUMMARY:
The main purpose is to study, in comparison to classic Home Nursing Care Services (SSIAD), the effect of reinforced Home Nursing Care Services (SSIAD) on the occurrence of hospitalizations

DETAILED DESCRIPTION:
It's a non-interventional, multi-centred, controlled study.

Inclusions will start with patients benefit from a so-called "reinforced" bed in the experimental Home Nursing Care Services (SSIAD), that is, with a score between 11 and 21 on the regional public health authorities (ARS) score. Patients from the classic Home Nursing Care Services SSIAD (control arm) will be inclused on a matching mode to the individual clinical profiles of patients recruited into the reinforced Home Nursing Care Services (SSIAD). Matching will be based on age, sex, and comorbidity score (Charlson scale). Screening for matching will be done by a geriatric physician appointed by the sponsor. Once screened in, patients will be proposed the study by the Home Nursing Care Services SSIAD lead investigator who provides home care. Patients in the control arm will also express no opposition. For each patient accepting the study, their family caregiver - if there is one - will also be proposed the study. Various data: Prescription medicinal, reason and duration of hospitalization, number and reason for emergency department presentations, independence and dependency scores and other scales will be collected retrospectively, at inlcusion (J0) , then monthly (M1 to M12).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years old
* Having obtained a place in SSIAD by medical prescription
* Able to understand and respond to study questionnaires and evaluations with or without the Assistance of a third party
* Resident in territories of activities of the SSIAD participating in assessment
* With social coverage
* Having expressed non-oppostion to his participation in study and documented in his medical file
* Only for patients in " einforced SSIAD ": patient with a so-called "reinforced" bed financed by " Regional Public Health authorities " (ARS) of Ile-de-France, and with a score between 11 and 21 on the ARS score

Exclusion Criteria:

* Age < 60 years old
* Expressing his opposition to participate in the study
* Not resident in the territory of activity of SSIAD
* Requires only technical care and management in the act
* Unable to understand and respond to study questionnaires and evaluations, even with third party assistance

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is elderly, polypathological patients who have been prescribed SSIAD. Patients eligible to participate in Reinforced SSIAD experiment are those who meet inclusion and non-inclusion criteria listed below. Patient selection will be done in the SSIAD themselves.
Sampling Method: Non-Probability Sample
Enrollment: 677 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of hospitalization frequency for patients with Reinforced SSIAD compared to similar patients in classic SSIAD. | 12 months
  Assess the hospitalization frequency for patients with an enhanced SSIAD placement compared to similar patients in conventional SSIAD.

SECONDARY OUTCOMES:
Assessment of commorbidity risk according Charlson score | 12 months
Assessment of the degree of patient dependence according "Index of Independence in Activities of Daily Living" KATZ scale | 12 months
Assessment of patient's level of dependence through an appreciation of instrumental activities of daily living according Lawton scale | 12 months
Assessment of teh degree of autonomy according AGGIR score | 12 months
Assessment of quality of life according "Nottingham health profile" scale | 12 months
Assessment of health-related quality of life according SF-36 (Medical outcome study Short-Form health survey-36 items) | 12 months
Assessment of the emotional, physical and financial burden on a caregiver according Zarit burden scale | 12 months
Assessment of qualityof life for caregiver according "36-Item Short Form Survey" (SF-36) Score | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- SSIAD SAPA, 139 Boulevard Saint-Denis, Courbevoie, Île-de-France Region, France